CLINICAL TRIAL: NCT00945906
Title: A Prospective, Multicenter, Open Enrollment Study of Human Plasma-Derived Factor XIII Concentrate in Subjects With Congenital Factor XIII Deficiency
Brief Title: An Open Enrollment Study of Factor XIII Concentrate in Subjects With Congenital Factor XIII Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BI71023_3002; 1488 (Other: CSL Behring)
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Factor XIII Deficiency
Keywords: Hereditary Factor XIII deficiency; Factor XIII
MeSH Terms: conditions — Factor XIII Deficiency | interventions — Factor XIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FXIII (Experimental): Subjects were administered FXIII Concentrate (Human) by intravenous (IV) infusion approximately every 28 days to maintain a trough FXIII level of approximately 5 to 20%.
  Interventions: Biological: FXIII Concentrate (Human) (FXIII)

INTERVENTIONS:
Biological: FXIII Concentrate (Human) (FXIII) — Doses will be guided by the individual subject's most recent FXIII activity levels, with the objective of dosing every 28 days to maintain a trough FXIII activity level of approximately 5 to 20%.
  Subjects enrolled in this study who have not received at least 3 doses of FXIII Concentrate in a previous study of this product (i.e., NCT00640289, NCT00885742, or NCT00883090) will initially receive a dose of 40 U/kg by intravenous (IV) infusion.
  Other Names: Fibrogammin-P®; Corifact®

SUMMARY:
Congenital deficiency of factor XIII is an extremely rare inherited disorder associated with potentially life-threatening bleeding. Factor XIII Concentrate is given to patients whose blood is lacking factor XIII. Factor XIII Concentrate works by assisting blood in the usual clotting process, thereby preventing bleeding.

In this study, patients will be treated with FXIII Concentrate (Human) and followed closely to determine that they receive the dose of FXIII Concentrate (Human) that will best minimize the chance of bruising and bleeding. The purpose of the study is to provide FXIII Concentrate (Human) to patients until the product becomes commercially available in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent for study participation obtained before undergoing any study specific procedures
* Diagnosed with congenital FXIII deficiency requiring prophylactic treatment
* Males and females of any age

Exclusion Criteria:

* Diagnosis of acquired FXIII deficiency
* Administration of a FXIII-containing product, including blood transfusions or other blood products, within 3 weeks prior to the Baseline/Day 0 Visit
* Any known congenital or acquired coagulation disorder other than congenital FXIII deficiency
* Use of any other IMP within 4 weeks prior to Baseline/Day 0 Visit
* Female subjects of childbearing potential not using, or not willing to use, a medically reliable method of contraception for the entire duration of the study
* Suspected inability (e.g., language problems) or unwillingness to comply with study procedures or history of noncompliance
* Any laboratory finding or medical condition which, in the opinion of the Investigator, would put the subject or subject's disease management at risk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (25):
- United States (25):
  - Study Site, Dothan, Alabama
  - Study Site, Oakland, California
  - Study Site, Orange, California
  - Study Site, San Francisco, California
  - Study Site, Stockton, California
  - Study Site, Fort Myers, Florida
  - Study Site, Miami, Florida
  - Study Site, St. Petersburg, Florida
  - Study Site, New Orleans, Louisiana
  - Study Site, Boston, Massachusetts
  - Study Site, Ann Arbor, Michigan
  - Study Site, Detroit, Michigan
  - Study Site, Kansas City, Missouri
  - Study Site, Las Vegas, Nevada
  - Study Site, Lebanon, New Hampshire
  - Study Site, Albany, New York
  - Study Site, New York, New York
  - Study Site, Chapel Hill, North Carolina
  - Study Site, Columbus, Ohio
  - Study Site, Hershey, Pennsylvania
  - Study Site, Sioux Falls, South Dakota
  - Study Site, Nashville, Tennessee
  - Study Site, Dallas, Texas
  - Study Site, Houston, Texas
  - Study site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FXIII
Started | 61
Completed | 54
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Did not want to return for last visit | 2
Not completed — Unable to return for last visit | 2
Not completed — Moved to another country | 2

BASELINE CHARACTERISTICS:
Arm/Group | FXIII
Number analyzed (Participants) | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 18.5 (12.48)
Age, Customized [Number; unit: participants]
  < 16 years | 29
  16 to < 65 years | 32
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of subjects with any treatment-emergent adverse event (AE), treatment-related AE or serious AE (SAE). Treatment-related AEs are defined as AEs whose relationship to treatment is related, or possibly related and AEs with missing relationship.
Time Frame: After the first infusion until study completion. Study completion is up to 2 years or until Factor XIII Concentrate (Human) is commercially available in the USA.
Population: The Safety Population consisted of all subjects who received a dose of Factor XIII Concentrate (Human) during the study. Treatment related AEs are events whose relationship to study treatment is related, or possibly related, in the opinion of the investigator. AEs with missing relationship are considered related to treatment.
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 61
participants
  Any treatment-emergent AE | 42
  Treatment-emergent and related AE | 2
  Serious AE | 2

2. Secondary Outcome: Hematology and Chemistry Testing
Description: Number of participants with treatment-emergent clinically significant hematology and/or chemistry laboratory parameter values.
Time Frame: After the first infusion and at the end-of-study (or withdrawal) visit.
Population: The Safety Population consisted of all subjects who received a dose of Factor XIII Concentrate (Human) during the study.
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 61
participants
  Clinically significant hematology test result | 1
  Clinically significant chemistry test result | 1

3. Secondary Outcome: FXIII Antibody Testing
Description: Number of participants with serum Factor XIII antibodies.
Time Frame: Before the first infusion, then every 48 weeks, at the end-of-study (or withdrawal) visit and after a bleeding episode requiring treatment with a Factor XIII -containing product.
Population: The Safety Population consisted of all subjects who received a dose of Factor XIII Concentrate (Human) during the study.
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 61
participants
  Subjects with Factor XIII antibodies | 1
  Subjects without Factor XIII antibodies | 60

4. Secondary Outcome: FXIII Concentration
Description: Trough Factor XIII concentration.
Time Frame: Before the first infusion, at 24 and 48 weeks after the first infusion, and at the end-of-study (or withdrawal) visit.
Population: The Safety Population consisted of all subjects who received a dose of Factor XIII Concentrate (Human) during the study.
Measure: Mean (Standard Deviation); unit: Units/mL
Arm/Group | FXIII
Number analyzed (Participants) | 61
Units/mL
  Baseline (n = 35) | 0.0987 (0.03695)
  Week 4 (n = 28) | 0.1177 (0.03484)
  Week 8 (n = 8) | 0.1238 (0.02973)
  Week 12 (n = 8) | 0.1075 (0.03196)
  Week 16 (n = 4) | 0.1025 (0.04573)
  Week 20 (n = 5) | 0.1160 (0.03578)
  Week 24 (n = 41) | 0.1341 (0.03346)
  Week 28 (n = 3) | 0.1667 (0.06658)
  Week 32 (n = 2) | 0.0950 (0.02121)
  Week 36 (n = 3) | 0.1083 (0.07489)
  Week 40 (n = 3) | 0.0933 (0.04509)
  Week 44 (n = 1) | 0.0500 (0)
  Week 48 (n = 13) | 0.1246 (0.02961)
  Week 72 (n = 2) | 0.1400 (0.01414)

5. Secondary Outcome: Number of Subjects With at Least One Bleeding Episode
Description: Number of subjects with at least one bleeding episode at any time after the first infusion in the study, and the number of subjects with at least one bleeding episode requiring Factor XIII treatment.
Time Frame: as for outcome 1
Population: The Safety Population consisted of all subjects who received a dose of Factor XIII Concentrate (Human) during the study.
Measure: Number; unit: participants
Arm/Group | FXIII
Number analyzed (Participants) | 61
participants
  At least one bleeding episode (after treatment) | 10
  At least one bleeding episode requiring treatment | 1

6. Secondary Outcome: Number of Bleeding Episodes
Description: Number of bleeding episodes at any time after the first infusion in the study.
Time Frame: as for outcome 1
Population: The Safety Population consisted of all subjects who received a dose of Factor XIII Concentrate (Human) during the study.
Measure: Number; unit: Episodes
Arm/Group | FXIII
Number analyzed (Participants) | 61
Episodes | 14

ADVERSE EVENTS:
Time Frame: After the first infusion until study completion. Study completion is up to 2 years or until Factor XIII Concentrate (Human) is commercially available in the USA.
Description: The Safety Population consisted of all subjects who received a dose of Factor XIII Concentrate (Human) during the study.
Arm/Group | FXIII
Serious Adverse Events (participants affected / at risk) | 2/61
Other Adverse Events (participants affected / at risk) | 19/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FXIII (N=61)
Factor XIII inhibition (Blood and lymphatic system disorders) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FXIII (N=61)
Upper respiratory infection (Infections and infestations) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fever (General disorders) | 6 (7)
Bruising (Injury, poisoning and procedural complications) | 4 (5)
Vomiting (Gastrointestinal disorders) | 3 (4)
Headache (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.